CLINICAL TRIAL: NCT00296127
Title: A Relative Bioavailability Study Of Celecoxib Administered As Capsule Contents Sprinkled On Applesauce In Healthy Adult Volunteers
Brief Title: Study of Celecoxib Bioavailability in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A3191202
Record Dates: First submitted 2006-02-22; First posted 2006-02-24 (Estimated); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Celecoxib

INTERVENTIONS:
Drug: Celecoxib

SUMMARY:
To evaluate the bioavailability of celecoxib administered as capsule contents sprinkled onto applesauce relative to intact capsule

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects

Exclusion Criteria:

* Standard criteria for healthy volunteer studies

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24
Dates: Start 2006-02; Study Completion 2006-03

PRIMARY OUTCOMES:
Relative bioavailability of celecoxib administered as capsule contents sprinkled onto applesauce relative intact capsule after a single dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3191202&StudyName=Study+of+celecoxib+bioavailability+in+healthy+subjects+